CLINICAL TRIAL: NCT03414346
Title: Comparisons of Differents Percentages of Water Effectiveness During Cryotherapy Application in Reducing Superficial Skin Temperature: A Randomized Single-blind Clinical Trial.
Brief Title: Analysis of the Effects on Human Tissues After Application of Therapeutic Modalities.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alessandro Haupenthal (Other)
Collaborators: Santa Catarina Federal University (Other)
Responsible Party: Sponsor-Investigator, Alessandro Haupenthal, Principal Investigator, Universidade Federal de Santa Catarina
Organization: Universidade Federal de Santa Catarina (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1771454
Record Dates: First submitted 2017-10-31; First posted 2018-01-29 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Humans; Young Adults; Health
Keywords: Cryotherapy; Skin temperature; Physical therapy modalities; Physical therapy; Thermography; Pain measurement
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: A randomized single blind, crossover experimental study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exclusively ice pack: (Experimental): Ice pack application: 500 grams of crushed ice.
  Interventions: Other: Exclusively ice pack
- Ice pack added 10% of water: (Experimental): Wetted ice pack application: 500 grams of crushed ice added to 50 mL of water at room temperature.
  Interventions: Other: Ice pack added 10% of water
- Ice pack added 100% of water: (Experimental): Wetted ice pack application: 500 grams of crushed ice added to 500 mL of water at room temperature.
  Interventions: Other: Ice pack added 100% of water

INTERVENTIONS:
Other: Exclusively ice pack — Each subject will receive an experimental intervention of exclusively 500 grams of crushed ice. The intervention will last 20 minutes, and the order of application, expressed in % of water X ice, will be according to the randomization (realized in the first day). The pack will be wrapped in a band for improvement of the contac area. The subject will be asked to mark his pain level on the visual analogue scale (no pain score of 0 and pain as bad as it could be score of 10) every minute until the total time of the intervention.
  Arms: Exclusively ice pack:
Other: Ice pack added 10% of water — Each subject will receive an experimental intervention of ice pack added to 50 mL of water. The intervention will last 20 minutes, and the order of application, expressed in % of water X ice, will be according to the randomization (realized in the first day). The pack will be wrapped in a band for improvement of the contac area. The subject will be asked to mark his pain level on the visual analogue scale (no pain score of 0 and pain as bad as it could be score of 10) every minute until the total time of the intervention.
  Arms: Ice pack added 10% of water:
Other: Ice pack added 100% of water — Each subject will receive an experimental intervention of ice pack added to 500 mL of water. The intervention will last 20 minutes, and the order of application, expressed in % of water X ice, will be according to the randomization (realized in the first day). The pack will be wrapped in a band for improvement of the contac area. The subject will be asked to mark his pain level on the visual analogue scale (no pain score of 0 and pain as bad as it could be score of 10) every minute until the total time of the intervention.
  Arms: Ice pack added 100% of water:

SUMMARY:
As a therapeutic modality, cryotherapy is highly used for soft tissue damage control during acute and subacute stages. Cryotherapy is able to reduce pain, inflammatory condition, muscle spasm, nerve conduction, metabolic rate, edema formation and to prevent secondary hypoxic injury. These effects are due to the heat conduction, passing from tissue to different cryotherapy modalities, leading to tissue temperature reduction.

The diversity of cryotherapy modalities in clinical practice, like crushed-ice packs, frozen food, gel packs and wetted ice packs, are widely explored by studies. To achieve anesthesia by cryotherapy it's settled that the skin temperature must reach 13,6 degrees celsius (ºC). Ice packs are the most effective modality of cryotherapy when placed directly on the skin, this effectiveness is accentuated when ice packs are associated with water. To improve the contact area the pack must be wrapped.

Even though wetted ice packs are the most effective modality, there are few studies approaching it. There aren't studies analyzing an ideal percentage of water to ice in this modality either. Also, it isn't observed if the amount of water interferes on the conduction of the heat from the skin to the ice pack, and in rewarming time. Besides neither of the studies measures the amount of pain during cryotherapy application, and if there was any difference between wetted ice packs, and ice packs isolated.

Therefore, the purpose of this study is to analyze the most effective cryotherapy modality for reducing skin temperature, rewarming time, and the amount of discomfort during the application.

DETAILED DESCRIPTION:
The data for the sample size calculation was taken from Kanlayanaphotpron and Janwantanakul (2005), that also approached the cryotherapy application. The software used to calculate the sample was GPower 3.1.9.2. A 16 subjects sample were obtained to reach a power of 90%, needed to detect a difference on the average of the groups in repeated measures with an alpha of 5%. The subjects will be chosen through social media and informal invitations.

The subjects will attend to the laboratory four times, the first day for orientation and measurements (body mass and skinfold), and the data collection will start on the second day.

The room temperature will be set between 23 ° C and 25 ° C, and the humidity around 70%. The subject will be in supine position on the stretcher, relaxed and instructed not to touch the right thigh region for 20 minutes before the intervention to stabilize the body temperature. The thigh will be measured and the center marked to determine the place where the pack will settle and the temperature collected.

The intervention will last 20 minutes, and the order of application will be according to the randomization. The subject will be asked to mark his pain level on the visual analogue scale every minute.

The temperature of the right thigh will be measured by infrared thermography, before the intervention, right after the removal and every minute until the total time of the intervention.

To summarize the data, it will be used descriptive statistics, the values of average, standard deviation and the collected measurements will be identified. Through Shapiro-Wilk test the distribution of data regarding normality will be verified. To compare the initial and the final test values the ANOVA and the post-hoc of Bonferroni will be used. In the case of data being out of the normal standards, a transformation will be used to reach the normality. If the data still don't reach the normality after the transformation, the non-parametric tests will be used (Mann-Whitney e Kruskal Walis). The confidence level adopted for all tests will be 95% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* No orthopedic injury in three months prior to the study;
* A minimum of 18 years of age, and a maximum of 40 years;
* Female;
* Must agree not to practice exercise the day before the study and not ingest caffeine, alcohol, or foods one hour before intervention.

Exclusion Criteria:

* Cold hypersensitivity and urticaria;
* Cold hyposensitivity;
* Raynaud's phenomenon diagnosed;
* Any thigh open wound;
* Muscular or neurological disease;
* Diabetes diagnosed;
* Cigarette smokers.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The most effective cryotherapy modality | 3 days
  Evaluation of the most effective percentage of water and ice, as a cryotherapy modality, in attenuating skin temperature. It will be evaluated in three visits, 24 hours apart each.

SECONDARY OUTCOMES:
Rewarming after ice application. | 3 days
  The skin temperature will be verified before the application of cryotherapy and after during 40 minutes, 2 minutes apart each measure.
Recurrence of pain. | 3 days
  The patient will be instructed to point the amount of pain minute by minute from time 0 to 20 minutes of application.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Haupenthal, Doctorate, Study Director — Santa Catarina Federal University
Locations (1):
- Santa Catarina Federal University, Araranguá, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belitsky RB, Odam SJ, Hubley-Kozey C. Evaluation of the effectiveness of wet ice, dry ice, and cryogenic packs in reducing skin temperature. Phys Ther. 1987 Jul;67(7):1080-4. doi: 10.1093/ptj/67.7.1080. PMID 3602101
- [Background] Chesterton LS, Foster NE, Ross L. Skin temperature response to cryotherapy. Arch Phys Med Rehabil. 2002 Apr;83(4):543-9. doi: 10.1053/apmr.2002.30926. PMID 11932859
- [Background] Dykstra JH, Hill HM, Miller MG, Cheatham CC, Michael TJ, Baker RJ. Comparisons of cubed ice, crushed ice, and wetted ice on intramuscular and surface temperature changes. J Athl Train. 2009 Mar-Apr;44(2):136-41. doi: 10.4085/1062-6050-44.2.136. PMID 19295957
- [Background] Enwemeka CS, Allen C, Avila P, Bina J, Konrade J, Munns S. Soft tissue thermodynamics before, during, and after cold pack therapy. Med Sci Sports Exerc. 2002 Jan;34(1):45-50. doi: 10.1097/00005768-200201000-00008. PMID 11782646
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Herrera E, Sandoval MC, Camargo DM, Salvini TF. Effect of walking and resting after three cryotherapy modalities on the recovery of sensory and motor nerve conduction velocity in healthy subjects. Rev Bras Fisioter. 2011 May-Jun;15(3):233-40. doi: 10.1590/s1413-35552011000300010. PMID 21829988
- [Background] Jutte LS, Merrick MA, Ingersoll CD, Edwards JE. The relationship between intramuscular temperature, skin temperature, and adipose thickness during cryotherapy and rewarming. Arch Phys Med Rehabil. 2001 Jun;82(6):845-50. doi: 10.1053/apmr.2001.23195. PMID 11387593
- [Background] Kanlayanaphotporn R, Janwantanakul P. Comparison of skin surface temperature during the application of various cryotherapy modalities. Arch Phys Med Rehabil. 2005 Jul;86(7):1411-5. doi: 10.1016/j.apmr.2004.11.034. PMID 16003673
- [Background] Oosterveld FG, Rasker JJ, Jacobs JW, Overmars HJ. The effect of local heat and cold therapy on the intraarticular and skin surface temperature of the knee. Arthritis Rheum. 1992 Feb;35(2):146-51. doi: 10.1002/art.1780350204. PMID 1734903
- [Derived] de Estefani D, Ruschel C, Beninca IL, Dos Santos Haupenthal DP, de Avelar NCP, Haupenthal A. Volume of water added to crushed ice affects the efficacy of cryotherapy: a randomised, single-blind, crossover trial. Physiotherapy. 2020 Jun;107:81-87. doi: 10.1016/j.physio.2019.12.005. Epub 2019 Dec 16. PMID 32026839